CLINICAL TRIAL: NCT02618330
Title: The Clinical Evaluation of Two Different Film Thicknesses of Clear Overlay Retainer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yafen Zhu (Other)
Responsible Party: Sponsor-Investigator, Yafen Zhu, PHD candidate, Sichuan University
Organization: Sichuan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: WCHSIRB-ST-2013-094
Record Dates: First submitted 2015-11-25; First posted 2015-12-01 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Retention
MeSH Terms: interventions — Orthodontic Retainers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- retainer: 0.75-mm-thick film (Experimental)
  Interventions: Device: retainer
- retainer: 1.00-mm-thick film (Experimental)
  Interventions: Device: retainer

INTERVENTIONS:
Device: retainer — 24 h wearing whether 0.75-mm-thick or 1.00-mm-thick film retainer

SUMMARY:
The aims of this study were to compare health related quality of life, comforts degrees，retention effectiveness, and failure rates as well as survival times between two clear overlay retainers with different thicknesses, thus to provide basis information regarding appropriate selections of the thickness of clear overlay retainers.

ELIGIBILITY:
Inclusion Criteria:

* Patients after active orthodontic treatment;
* Must be healthy without systemic and oral diseases;
* The central incisors, canines and first molars of both upper and lower arches must be existed;
* Agreed to the trial and signed informed consent forms, either by themselves, or their parents.

Exclusion Criteria:

* Oral habits such as bruxism and clenching,
* Do not accept this type of retainers

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Survival times via recording to the patients' re-visit | one year

SECONDARY OUTCOMES:
SF-36 scale for Quality of life | one month
Comfort degrees assessed through Visual Analog Score | one month
Retention effectiveness assessed according to 3D models | one year

REFERENCES:
- [Derived] Zhu Y, Lin J, Long H, Ye N, Huang R, Yang X, Jian F, Lai W. Comparison of survival time and comfort between 2 clear overlay retainers with different thicknesses: A pilot randomized controlled trial. Am J Orthod Dentofacial Orthop. 2017 Mar;151(3):433-439. doi: 10.1016/j.ajodo.2016.10.019. PMID 28257727